CLINICAL TRIAL: NCT01502943
Title: Studies of Traditional Chinese Medicine Clinical Efficacy Evaluation Index With Stable Angina Pectoris of Coronary Heart Disease as an Example
Brief Title: Studies of Traditional Chinese Medicine Clinical Efficacy Evaluation Index
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Liaoning University of Traditional Chinese Medicine (Other)
Collaborators: Ministry of Science and Technology of the People´s Republic of China (Other Government)
Responsible Party: Principal Investigator, YANG Guan-lin, Principal of Liaoning university of TCM, Liaoning University of Traditional Chinese Medicine
Allocation: Randomized | Model: Parallel | Masking: Triple
Other Study IDs: 2009ZX09502-029
Record Dates: First submitted 2011-12-15; First posted 2012-01-02 (Estimated); Last update posted 2012-01-02 (Estimated); Status verified 2011-12

CONDITIONS: Coronary Heart Disease; Stable Angina Pectoris
Keywords: Complementary Therapies; Traditional Chinese Medicine; Quality of life; Seattle angina questionnaire (SAQ); SF-12; Measure Your Medical Outcome Profile (MYMOP); Phlegm and blood stasis Syndrome; Qi deficiency and blood stasis Syndrome; Invigorating Spleen to Remove Phlegm or replenish Qi; Activating blood and dissolving stasis; Traditional Chinese medicine SYndrome Scale (TCMsys); Patients Report Outcomes(PRO); clinical efficacy; evaluative index
MeSH Terms: conditions — Coronary Disease; Angina, Stable | interventions — Long-Term Synaptic Depression; Atorvastatin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Phlegm and blood stasis Syndrome G (Experimental)
  Interventions: Drug: Louxiangdan Tongxin granules; Drug: Western basis treatment
- Phlegm and blood stasis control G (Placebo Comparator)
  Interventions: Drug: TCM granules placebo; Drug: Western basis treatment
- Qi deficiency and blood stasis G (Experimental)
  Interventions: Drug: Chixiangshen Tongxin granules; Drug: Western basis treatment
- Qi deficiency and blood stasis control G (Placebo Comparator)
  Interventions: Drug: TCM granule placebo plus western basis treatment; Drug: Western basis treatment

INTERVENTIONS:
Drug: Louxiangdan Tongxin granules — TCM treatment:
  Decoction: Louxiangdan Tongxin granules Herbs:Danshen 10g、Chenxiang 1g、Gualou10g、Xiebai 10g、Banxia6g、Chuanxiong 6g 、Dangshen 10g、Zhiqiao 6g、Taoren 10g、Guizhi 6g Therapeutic Principle:Invigorating Spleen to Remove Phlegm and activating blood and dissolving stasis, at least 6 kinds of TCM herbs can be chosen and their dosages be adjusted according to Syndrome Differentiation.
  Usage:Once 100ml, twice per day after breakfast and supper.
  Other Names: Louxiangdan Tongxin granules from Jiangyin Tianjiang Pharmaceutical Co., Ltd
  Arms: Phlegm and blood stasis Syndrome G
Drug: TCM granules placebo — Chinese medicine granules placebo: once 100ml, twice per day after breakfast and supper.
  Other Names: TCM placebo granules from Jiangyin Tianjiang Pharmaceutical Co., Ltd
  Arms: Phlegm and blood stasis control G
Drug: Chixiangshen Tongxin granules — TCM treatment:
  Decoction: Chixiangshen Tongxin granules Herbs: Chishao 10g, Chenxiang 1g, Danggui 10g, Jupi 10g, Yanhusuo 6g, Chuanxiong 6g, Dangshen 10g, Huangqi 6g, Taoren 10g, Honghua 10g Therapeutic Principle:Invigorating Spleen to Replenish Qi and activating blood and dissolving stasis, at least 6 kinds of TCM herbs can be chosen and their dosages be adjusted according to Syndrome Differentiation.
  Usage:Once 100ml, twice per day after breakfast and supper.
  Other Names: Chixiangshen Tongxin granules from Jiangyin Tianjiang Pharmaceutical Co., Ltd
  Arms: Qi deficiency and blood stasis G
Drug: TCM granule placebo plus western basis treatment — Chinese medicine granules placebo: once 100ml, twice per day after breakfast and supper.
  Other Names: TCM placebo granules from Jiangyin Tianjiang Pharmaceutical Co., Ltd
  Arms: Qi deficiency and blood stasis control G
Drug: Western basis treatment — Aspirin: 100mg pd. P.O.( patients who have Aspirin resistance or Allergy can replaced with Piece clopidogrel 75mg pd. P.O.) Atorvastatin calcium (Lipitor): 10mg pd. P.O.( patients who have Atorvastatin calcium resistance or Allergy can replaced with Additive amount of pravastatin equal to 10mg Lipitor) Nitroglycerin: sublingual necessary.
  Other Names: Aspirin from Liaoning WanLong medicine Co.,Ltd; Atorvastatin calcium (Lipitor) from Liaoning Pharmaceutical foreign trade corporation

SUMMARY:
The purpose of the trial is to take stable angina pectoris of coronary heart disease (CHD) as examples to build a standard evaluation system for efficacy of traditional Chinese medicine (TCM).

1. Studies of evaluating reliability, validity and reactivates of Patients Report Outcomes of CHD and self-administrated scale of Stable Angina Pectoris
2. research on all indicators of CHD, and analyze their characteristics, target and function
3. theory of Invigorating Spleen to Remove Phlegm or replenish Qi, and activating blood and dissolving stasis as an example for clinical efficacy evaluation.

DETAILED DESCRIPTION:
Clinical efficacy is the basis of traditional Chinese medicine development, and scientific evaluation of TCM clinical efficacy and its effectiveness is the way to push TCM modernized and international. TCM theories of Overall concept and Differentiation for life science and diseases are hard to be generally accepted. Besides, no unified and standard methods fit to evaluate the TCM clinical efficacy. Thus, there is a need to do a deeper research of methodology, evaluative index, and evaluative criteria in order to guide the evaluation of TCM clinical efficacy.

Based on the situation above, the study aims to choose the best and characteristic evaluative index of clinical efficacy, compare the demand among practitioners, patients and care givers. After data collected, a new cluster of index among Biochemical, patients report outcomes, endpoint indicators, and TCM soft indicators could be constituted and analyzed to use in respective way according to their characteristics, target and function.

ELIGIBILITY:
Inclusion criterion：

* The diagnosis standard according with stable angina coronary heart disease
* The participants with any one of the below six standards are included:

  * history of myocardial infarction previously
  * PCI postoperative patients
  * CT showing more than 50% coronary stenosis
  * Coronary angiography showing more than 50% coronary stenosis
  * positive results of the electrocardiogram
  * ischemia changes in the electrocardiogram recently
* The Patients with disease history more than three months, attacked in the recent one month
* Standard according to the phlegm and blood stasis syndrome or Qi deficiency and blood stasis syndrome of the traditional Chinese medicine
* Male: 45 years old < 75 years old
* Female: 50 years old < 75 years old
* Participants signed the agreement paper voluntarily.

Exclusion criterion:

* Participants with Acute coronary syndrome (ST segment elevation myocardial infarction, non ST segment elevation myocardial infarction, unstable angina), asymptomatic myocardial ischemia,ischemic cardiomyopathy,the myocardial infarction happening in the 3 months before the test
* Participants with rheumatism heart disease, hyper thyroid heart disease, hypertensive heart disease, myocarditis, cardiomyopathy
* Participants with Cervical disease, gallbladder cardiac syndrome, stomach and esophageal reflux, aortic dissection
* Participants with acute cerebral infarction and cerebral hemorrhage
* Participants with severe heart failure, lung function, liver function (AST, ALT 1.5 times normal standard), kidney function (BUN, Cr more than the normal standard), hematopoietic system and endocrine systems and serious primary disease, malignant tumor, gastrointestinal bleeding, gastric ulcer and are prone to bleed
* the Participants can not complete the whole test
* The serious high blood pressure and hard to control (SBP >= 180 mmHg or DBP >=110 mmHg)
* Participants of acute or chronic cardiac dysfunction with heart function III-IV
* Participants has been included in other clinical studies in one month;
* Participants with glaucoma
* Participants with Pregnancy Or Lactation ,Allergy
* Participants with mental disorder, or nervous disease, or illiteracy, or bad compliance for questionnaire

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 480 (Actual)
Dates: Start 2011-05; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
TCM characteristics evaluative index: Traditional Chinese medicine SYndrome Scale (TCMsys) (new developed） | Taken at day 1 (baseline) and Change from Baseline in 2nd,4th,8th week
New developed Quality of life evaluative index: patients report outcomes for SAP | Taken at expected day 7 in the screen period, day 1 (baseline) and Change from Baseline in 2nd,4th,8th week
New developed Quality of life evaluative index: self-administrated scale of SAP | Taken at expected day 7 in the screen period, day 1 (baseline) and Change from Baseline in 2nd,4th,8th week

SECONDARY OUTCOMES:
Symptoms evaluative index: Measure Your Medical Outcome Profile (MYMOP), Angina incentives, symptom score scale, rate of nitroglycerin, angina classification, heart function classification | Taken at day 1 (baseline) and Change from Baseline in 2nd,4th,8th week; and all except MYMOP taken one more at expected day 7 in screen
Biochemical index: ECG, ECG exercise test, blood lipids, blood glucose (fasting glucose), Blood, urine, liver function, renal function, coagulation, echocardiography (including heart function), coronary CT (some hospitals choose to do) | Taken at expected day 7 in the screening period (baseline) and Change from Baseline in 8th week
Quality of life evaluative index: Seattle angina questionnaire (SAQ) | Taken at day 1 (baseline) , Change from Baseline in 2nd, 4th, 8th, 12th week
Quality of life evaluative index: short form-12 (SF-12) | Taken at day 1 (baseline), Change from Baseline in 2nd, 4th, 8th, 12th week
TCM characteristics evaluative index: Traditional Chinese medicine Syndrome Scale 2 (criteria) | Taken at expected day 7 in the Screening period,and Change from Baseline in 2nd,4th,8th week
Endpoint index （Cardiovascular events, non-cardiovascular events, death, hospitalization due to coronary heart disease cases） | Taken at 2nd, 4th, 8th, 12th, 26th week

CONTACTS AND LOCATIONS:
Overall Officials: Guanlin Yang, Study Chair — Liaoning University of TCM
Locations (10):
- China (10):
  - Affiliated hospital of Changchun university of TCM, Changchun, Jilin
  - Jilin integrative Chinese and western medicine hospital, Changchun, Jilin
  - Dalian integrative of Chinese and Western medicine hospital, Dalian, Liaoning
  - Dandong TCM hospital, Dandong, Liaoning
  - Fuxin TCM hospital, Fuxin, Liaoning
  - Affiliated hospital of Liaoning university of TCM 2, Shenyang, Liaoning
  - Affiliated hospital of Liaoning university of TCM, Shenyang, Liaoning
  - Shengjing Hospital of China Medical University, Shenyang, Liaoning
  - Yingkou TCM hospital, Yingkou, Liaoning
  - Affiliated hospital of Tianjin university of TCM, Tianjin, Tianjin Municipality